CLINICAL TRIAL: NCT02749708
Title: Phase I/II Study of IRX5183 in Relapsed and Refractory Acute Myeloid Leukemia (AML) and High Risk Myelodysplastic Syndrome (MDS)
Brief Title: Study of IRX5183 in Relapsed and Refractory Acute Myeloid Leukemia and High Risk Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study drug supply expired and could not be renewed.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Io Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J15219; IRB00083855 (Other: JHMIRB)
Record Dates: First submitted 2016-04-05; First posted 2016-04-25 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS); Chronic Myelomonocytic Leukemia (CMML)
Keywords: IRX5183; relapsed/refractory AML; high-risk MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose level 1 (Experimental): IRX5183 50 mg daily
  Interventions: Drug: IRX5183
- Dose level 2 (Experimental): IRX5183 75 mg daily
  Interventions: Drug: IRX5183

INTERVENTIONS:
Drug: IRX5183 — IRX5183 will be administered orally daily on days 1-28 of each cycle for 2 cycles of induction. In the phase I part of the study, there will be 3 dose levels (dose level 1 [DL1] with 50 mg, DL2 with 75 mg, and DL3 with 100 mg), with 1 additional dose level to be only used if excessive toxicity noted at the DL1. There will be no intra-patient dose escalation. A phase II portion of the study was originally planned, but the study was terminated prior to phase II enrollment.

SUMMARY:
The purpose of this study is to evaluate the use of IRX5183 in 1) patients with relapsed and/or refractory AML and 2) patients with high-risk MDS or chronic myelomonocytic leukemia (CMML).

DETAILED DESCRIPTION:
This research is being done to learn about the safety and effectiveness of an investigational drug, IRX5183, in treating acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS). IRX5183 is a derivative of Vitamin A. IRX5183 is a drug that is designed to cause cancer cells to mature and then die. It is thought that it will stop the uncontrolled growth of leukemia cells.

These are 2 parts to this study. The purpose of the first part is to test the safety of IRX5183 at different dose levels. The investigators want to find out what effects, good and/or bad, it has on AML or MDS. Once the investigators figure out the best and safest dose of IRX5183, the investigators will enter the second part of the study using this dose. The purpose of the second part is to see if IRX5183 is effective as a treatment for AML or MDS. To date, IRX5183 has been used in about 25 people.

The first part of the study is called a "Phase I" study. Phase I studies use drugs starting at low doses and slowly increase the amounts of the study drugs that are given to people until the side effects of the drugs are too high to give more. This means that not all people in the study will get the same dose of IRX5183. Doses at the beginning of the study will be lower than doses at the end of the study. Because of the design of the study, some people may get doses that are too low to have an effect, and other people will probably get doses that cause side effects.

People with AML, MDS, or CMML that has 1) not responded to standard therapy or 2) has returned after a previous response may join.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand and voluntarily sign an informed consent form.
2. Age ≥ 18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Pathologically confirmed disease with A or B as follows:

   A) AML patients who either have:
   * Relapsed or refractory disease after receiving one or more courses of induction chemotherapy, hypomethylating agent therapy, or bone marrow transplant or
   * de novo AML but not deemed to be a candidate for conventional therapy based on age, co-morbidities, or patient preference

   B) MDS, CMML, or MDS/myeloproliferative neoplasm (MPN) with high risk features as defined below who have relapsed after initial response or are refractory (failure to achieve a complete remission (CR), partial remission (PR), or hematologic improvement (HI)) after receiving at least 4 cycles of hypomethylating agents 5-azacitidine or decitabine ± other therapies ± bone marrow transplant OR with de novo MDS but have refused to receive hypomethylating therapy:
   * Intermediate (INT)-2 or high International Prognostic Scoring System (IPSS) score OR high or very high revised IPSS (IPSS-R) or
   * Secondary MDS (defined as MDS developing in a patient with an antecedent hematologic disorder or any patient with prior chemotherapy or radiation exposure) or
   * INT-1 IPSS or intermediate IPSS-R MDS with excess blasts (≥5% blasts in bone marrow) or transfusion-dependency or
   * MDS progressing to oligoblastic AML with 21-30% bone marrow blasts or
   * CMML or MDS/MPN with ≥ 5% marrow blasts, transfusion-dependency, abnormal karyotype, or proliferative features (white blood cell count ≥13,000/µL, splenomegaly on physical examination, or extramedullary disease)
5. Eastern Cooperative Oncology Group performance status of ≤ 2 at study entry or Karnofsky > 60%.
6. Laboratory test results within these ranges:

   Creatinine level of 3 mg/dL or lower, total bilirubin ≤ 3 mg/dL unless due to Gilbert's syndrome, hemolysis, or ineffective hematopoiesis, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x upper limit of normal, white blood count (WBC) ≤ 10,000/µL
7. Patients must not have received any other treatment for their disease, including hematopoietic growth factors, aside from hydroxyurea for count control, within three weeks of beginning the trial, and should have recovered from all toxicities of prior therapy (to grade 0 or 1).
8. Patients requiring hydroxyurea to bring WBC below 10,000/µL prior to study enrollment will require a 48-hour washout prior to starting the study drug.
9. Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to start of IRX5183.
10. Patients must have no clinical evidence of central nervous system (CNS) or pulmonary leukostasis, disseminated intravascular coagulation, or CNS leukemia.

Exclusion Criteria:

1. Any serious medical condition or uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, laboratory abnormality, or psychiatric illness/social situations that would limit compliance with study requirements or prevent the subject from signing the informed consent form.
2. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
3. Use of any other experimental drug or therapy within 21 days of baseline.
4. Known hypersensitivity or history of allergic reactions attributed to compounds of similar chemical or biologic composition to IRX5183.
5. Prior use of other retinoid therapies in the 3 months prior to enrollment in the study.
6. Patients with other active cancers receiving anti-cancer agents, with exceptions being hormonal therapy for breast or prostate cancer and skin cancers treated with local therapies only.
7. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier (e.g. alopecia, hypothyroid, neuropathy, etc.).
8. Pregnant women are excluded from this study because of potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with IRX5183, breastfeeding should be discontinued if the mother is treated with IRX5183.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and tolerability of IRX5183 in phase I using National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0, to determine dose limiting toxicities (DLTs) and the recommended phase 2 dose (RP2D). | 2 years
  We will determine DLTs at specified dose levels to determine the RP2D.
Determine the best overall response rate (ORR) per International Working Group (IWG) criteria with the RP2D after at least 2 therapy cycles. | 2 years
  The primary endpoint of phase II is best ORR per IWG criteria after at least 2 cycles of therapy. If enough patients achieve an objective response, enrollment will continue to a second stage, per a Simon's 2 stage design.

SECONDARY OUTCOMES:
Measure trough plasma levels of IRX5183 on day 1 and day 14. | 4 years
  To determine pharmacokinetic (PK) parameters of IRX5183, we will obtain trough peripheral blood samples during the first cycle of therapy.
Measure peak plasma/bone marrow levels of IRX5183 on day 1 and day 14. | 4 years
  To determine PK parameters of IRX5183, we will obtain peak peripheral blood/bone marrow samples during the first cycle of therapy.
Determine flow markers of differentiation in the peripheral blood and/or bone marrow. | 4 years
Determine changes in cytogenetics in the peripheral blood and bone marrow before and after treatment with IRX5183. | 4 years
Determine the time to first and best response, per IWG criteria. | 4 years
Determine changes in transfusion requirements following therapy with IRX5183. | 4 years
Assess quality of life with the Functional Assessment of Cancer Therapy-leukemia (FACT-leu) questionnaire at baseline, after 2 cycles, and after 6 cycles of therapy. | 4 years
Determine event-free survival (EFS) for patients treated with IRX5183. | 4 years
Determine overall survival (OS) for patients treated with IRX5183. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Smith, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ambinder AJ, Norsworthy K, Hernandez D, Palau L, Paun B, Duffield A, Chandraratna R, Sanders M, Varadhan R, Jones RJ, Douglas Smith B, Ghiaur G. A Phase 1 Study of IRX195183, a RARalpha-Selective CYP26 Resistant Retinoid, in Patients With Relapsed or Refractory AML. Front Oncol. 2020 Oct 23;10:587062. doi: 10.3389/fonc.2020.587062. eCollection 2020. PMID 33194741

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT02749708/Prot_SAP_000.pdf